CLINICAL TRIAL: NCT00694811
Title: Liquid Very-Low-Energy Diets (VLEDs) in Obesity Treatment. Effects of Re-Feeding Duration On Weight Maintenance, Eating Behaviour and Health-Related Quality of Life
Brief Title: Effects of Re-Feeding Duration on Weight Maintenance After Weight Loss With Very-Low-Energy Diets (VLEDs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Lena Gripeteg, registered dietician, postgraduate student, Sahlgrenska University Hospital, Sahlgrenska Academy, University of Gothenburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUREG-1942
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Diet; Very-low-energy diet; Predictive factors; Re-feeding
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 1 week of re-feeding
  Interventions: Behavioral: Re-feeding duration
- B (Experimental): 6 weeks of re-feeding
  Interventions: Behavioral: Re-feeding duration

INTERVENTIONS:
Behavioral: Re-feeding duration — 1 or 6 weeks of re-feeding after VLED-induced weight loss
  Other Names: Dietary advice

SUMMARY:
The primary objective of the study is to test the hypothesis that prolonged re-feeding after VLED induced weight loss improves weight maintenance and eating behaviour

DETAILED DESCRIPTION:
VLED program:

During the initial 12 weeks, patients were encouraged to follow a strict liquid very-low-energy diet (470-820 kcal). They selected and paid themselves for one of the following commercially available diets; Modifast® (820 kcal), Nutrilett® (560 kcal) or Cambridgekuren® (470 kcal). Free consumption of non-caloric drinks (<6 kcal/100 g) was allowed. All patients had scheduled nurse visits at week 0 (baseline), 2, 5, 8, and 12. Body weight was registered at each visit and patients were given support and counselling to enhance VLED compliance. Side effects were monitored and a more frequent contact was offered if needed. All patients were encouraged to be physically active.

Dietary treatment:

Following VLED, dietary treatment advice was given during individual dietician counseling at nine study visits (week 12, 15, 18, 21, 26, 32, 38, 44, and 52). At week 12, the dietician assigned patients with ≥10% weight loss to treatment group according to randomization. Standardized written and oral instructions for one or six week re-feeding were provided; hence, participants as well as study staff were aware of group assignment. During re-feeding, ordinary meals were gradually re-introduced and VLED portions removed. Patients with one week re-feeding (Group 1) (instructed at week 12) started with breakfast for three days, added lunch (or dinner) the next four days, and thereafter the third meal was re-introduced and VLED discontinued. Patients with six week re-feeding (Group 6) (instructed at week 12, 15, and 18) started with one regular meal (patient's choice) for three weeks. A second meal was added the next three weeks, and at week eight the third meal was re-introduced and VLED discontinued. For both groups between-meal snacks (e.g. fruit) were recommended from the completion of the re-feeding periods.

Recommended energy intake was based on an estimated energy requirement minus 30% to achieve an energy-reduced level. Energy requirement was calculated from the equation of Harris-Benedict for estimation of basal metabolic rate, adjusted by factor 1.3 for total energy expenditure (moderate level of physical activity). Recommended energy distribution for breakfast, lunch and dinner was 20, 35 and 35% of daily energy intake, and 10% from snacks. Dietary prescriptions followed the Swedish Nutrition Recommendations. All patients were encouraged to increase their level of physical activity.

Power calculation and randomization:

Sample size calculations were based on data from a similar study. A sample size of 75 patients per treatment arm was derived, assuming 80% power to detect a 4 kg weight loss difference, SD 7 kg, statistical significance level P<0.05, and 35% dropout between week 12 and 52.

Two-hundred and sixty-nine patients started on the VLED regimen, and were after 12 weeks eligible for randomization if they had lost ≥10% of initial body weight. The randomization was stratified by the combination of sex and degree of weight loss (strictly greater than or less than 17.1% weight loss). Eligible patients were randomly assigned within each of the four strata to one of the two treatments (one or six weeks re-feeding) in blocks of size two, with equal allocation of treatments within each block. The randomization list was generated with a pseudo-random number generator, so that the resulting treatment sequence was reproducible and unpredictable.

The treatment allocation order was arranged in numbered, sealed envelopes and kept in separate boxes for each strata. At patient assignment, the envelope next in order was drawn from the appropriate strata box.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* BMI > 30 kg/m2
* speaking swedish

Exclusion Criteria:

* eating disorder
* unstable diabetes type 1
* unstable cardiac disease
* severe psychiatric disorder
* pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Weight development | 52 weeks

SECONDARY OUTCOMES:
Eating behaviour (Three Factor Eating Questionnaire) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Stenlöf, MD, Study Chair — Institute of Medicine, Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden